CLINICAL TRIAL: NCT05618886
Title: The Effect of Pelvic Floor Muscle Training for Urinary Incontinence in Nepalese Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bimika Khadgi, PT, Associate Professor, PhD candidate, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUSMS PT (WH)
Record Dates: First submitted 2022-10-31; First posted 2022-11-16 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Urinary Incontinence
Keywords: Nepali women, PFMT, intervention study
MeSH Terms: conditions — Urinary Incontinence | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The participants will be randomize into either education only (group A) or education plus PFMT (group B) 1:1 by concealed allocation (sealed envelope with A and B). After allocation, the participants will stay in their assigned intervention group for 1 year
Who Masked: Outcomes Assessor
Masking Description: A research assistant(assessor) will use a Samsung tablet with open data kit software to collect and record baseline questionnaire data containing socio-demographic variables and questions related to knowledge of UI (describe UI, the causes and treatment options and how participant's learnt about it), PFM and experience with PFMT of all the subjects. Assessor will not have any idea about the participant's in the treatment group and the control group. Assessor will be assessing through the patient reported questionnaire tool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Education given to all participants included before randomization. Information about UI, PFM and PFMT, together with lifestyle advices such as using the 'knack' (pre-contracting the PFM before coughing and sneezing), maintaining healthy weight, toilet habits, and reducing constipation and intra-abdominal pressure. The education session will last 30 minutes, and include a video (https://www.youtube.com/watch?v=XsDpfq10JMI) and a leaflet containing the information given.
  Interventions: Other: Education
- intervention group (Experimental): Along with education session, twelve weekly face-to-face sessions of PFMT with exercises individually or in groups with the women's health physiotherapist will be offered. PFMT will be taught on the basis of observation, vaginal palpation and camtech manometry, and will be individualized initially to suit each participant's ability within a protocol encouraging 10 close-to-maximum contractions and 6-8-second hold with a 10-second rest between contractions. During the first two appointments, participant will be instructed to perform two sessions with rest in between and thereafter three times 10 contractions if possible during each visit. The participants will be encouraged to perform daily PFMT (10 contraction x 3 10times, 3 sets) at home and will be asked to record their PFMT in an exercise diary
  Interventions: Other: Education and PFMT

INTERVENTIONS:
Other: Education — The education about urinary incontinence, PFM and PFMT together with lifestyle behavior modifications such as using the knack, maintaining healthy weight, toilet habits, and reducing constipation and intra-abdominal pressure will be provided along with the PFMT instruction.
  Arms: control group
Other: Education and PFMT — Along with education twelve weekly face-to-face sessions of PFMT with exercises individually or in groups with the women's health physiotherapist will be offered. PFMT will be taught on the basis of observation, vaginal palpation and camtech manometry, and will be individualized initially to suit each participant's ability within a protocol encouraging 10 close-to-maximum contractions and 6-8-second hold with a 10-second rest between contractions. During the first two appointments, participant's will be instructed to perform two sessions with rest in between and thereafter three times 10 contractions if possible during each visit. The participant's will be encouraged to perform daily PFMT (10 contraction x 3 10times, 3 sets) at home and will be asked to record their PFMT in an exercise diary.
  Arms: intervention group

SUMMARY:
The purpose of the study is to find the effectiveness of Pelvic floor muscle training (PFMT) for urinary incontinence (UI) among Nepalese women. After screening the women who meet the inclusion criteria will be included. Verbal and written consent will be taken from individual participants then the baseline questionnaire data containing socio-demographic variables and questions related to knowledge of UI, PFM and experience with PFMT and ICIQ UI SF will be collected. Then, a women's health physiotherapist will provide education about UI, PFM, PFMT and lifestyle advice. After the education session the randomisation of the participants into either education only (group A) or education plus PFMT (group B) 1:1 by concealed allocation (sealed envelope with A and B). After allocation, the participants will stay in their assigned intervention group for 1 year. After 12 weeks of the supervised intervention again ICIQ UI SF will be administered by a research assistant to both groups. In the 6th month again ICIQ UI SF will be administered by a research assistant to both groups. Finally, in the 12th month again ICIQ UI SF along with self-efficacy and knowledge questions will be assessed to find the effectiveness of the intervention. This data will help in the further development of the protocol or guideline for the Nepalese women.

DETAILED DESCRIPTION:
Urinary Incontinence (UI) is a widespread condition among women of all ages. UI is defined as involuntary urine leakage and categorized into three subcategories; the most common type Stress UI (SUI) concerns urine leakage associated with physical exertion, coughing and sneezing; Urge UI (UUI) involves a sudden urge to pass urine which is preceded or accompanied by urine leakage while mixed UI involves both SUI and UUI. UI has a negative impact on quality of life. It can cause social problems by creating embarrassment and negative self-perception, can reduce social interaction and physical activities, and also affect sexual relationship leading to anxiety and depression.

Population studies from numerous countries have reported that the prevalence of UI ranges from approximately 5%-70%, with most studies reporting a prevalence of UI to be between 25-45%. Few studies have examined UI in Nepal. One study among women with gynecological disorders in eastern Nepal reported a prevalence of UI to be as high as 50%. A large community based survey among 14,469 women in rural Nepal, found the prevalence of SUI and UUI to be 24% and 14%, respectively.

The large variation of prevalence between studies could be because of methodological differences, such as different data collection procedures with use of different questionnaires. The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is however the recommended subjective measure of severity of urinary loss and quality of life for those with UI. The questionnaire has been used in many studies for the assessment of UI and is available in different languages with good reliability and validity. So far, there is a lack of a Nepali version of the ICIQ-UI SF. Hence, it is a need to translate and cross-culturally adapt the ICIQ-UI SF into Nepali.

A recent Cochrane review showed that pelvic floor muscle training (PFMT) is effective for women with SUI, UUI, or mixed UI and is recommended as a first line conservative treatment over at least 3 months duration. The efficacy of PFMT is well established in national and international guidelines but to our knowledge no previous studies have assessed the effectiveness of PFMT for UI among Nepalese women.

ELIGIBILITY:
Inclusion Criteria:

* Between age of 18-45 years
* ICIQ grading above 3
* Understand Nepali language
* Willing to be included in the study
* Phone availability

Exclusion Criteria:

* Pregnant
* Planning for pregnancy within a 6 months period
* Waiting for gynaecological surgery
* History of bladder, renal, or uterine cancer
* Menopause
* Stage IV pelvic organ prolapse
* Cognitive or mental disorders
* Illness to mother or family members, not making exercising possible

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with UI
Enrollment: 136 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) will be used as primary outcome tool as it is recommended as self-reported patient outcome measure for UI. | Baseline, 12 week , 6month,12 month
  The ICIQ-UI SF consists of four items which evaluate the frequency, amount of leakage, overall impact of UI and self-diagnostic item. The overall score ranges from 0 to 21, with greater values indicating increased severity. The difference in change from baseline of ICIQ-UI SF scores of patients after intervention will report the effect of the intervention.

SECONDARY OUTCOMES:
Self-Efficacy Scale for Practicing Pelvic Floor muscle Exercise (SESPPFE) will be used to measure the self efficacy of PFMT as it is a valid and reliable outcome tool . | Baseline, 12 weeks, 6 months, 12 months
  SESPPFE is 17 items tool to measure self-efficacy of practicing PFM exercises with two components: self-efficacy score of 13 and outcome expectation score of 4. The interpretation will be done as higher scores means better self-efficacy or outcome expectation. The scores higher than 70% will be interpreted as relatively good self-efficacy.
The presence of contraction will be determined through the Rating Scale of contraction and also with A manometer from Camtech AS (Norway) | Baseline,12 weeks
  To ensure valid measurements, only PFM contractions with simultaneous visible inward movement of the perineum and a manometer will be used. Through the manometer resting tone will be calculated as the difference between atmospheric pressure and the mean vaginal pressure at rest before and between the PFM contractions (cmH2O). Maximum volumetric contraction (MVC) will be calculated as a mean of three MVCs (cmH2O). PFM endurance will be recorded as a sustained maximal contraction for 10 seconds, quantified as the area under the curve (cmH2Osec)

OTHER OUTCOMES:
Baseline and knowledge questionnaire | baseline, 12months
  The baseline questionnaire will be containing socio-demographic variables and questions related to knowledge of UI PFM and experience with PFMT will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjeeta Acharya, PhD, Principal Investigator — KUSMS; Britt Stuge, PhD, Study Director — Oslo; Corlia Brandt, Study Director — WITS
Locations (2):
- Nepal (2):
  - Dhulikhel Hospital, Dhulikhel, Kavrepalanchok District- 3
  - Bimika Khadgi, Kathmandu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shijagurumayum Acharya R, Tveter AT, Grotle M, Khadgi B, Braekken IH, Stuge B. Pelvic floor muscle training programme in pregnant Nepalese women-a feasibility study. Int Urogynecol J. 2020 Aug;31(8):1609-1619. doi: 10.1007/s00192-019-04053-1. Epub 2019 Jul 25. PMID 31346671
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322